CLINICAL TRIAL: NCT00498485
Title: Phase IV - A Trial of Xyrem in the Treatment of Chronic Fatigue Syndrome.
Brief Title: Use of Xyrem to Improve Sleep in Chronic Fatigue Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawal of support.
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120060315
Record Dates: First submitted 2007-07-02; First posted 2007-07-10 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Fatigue Syndrome
Keywords: chronic; fatigue; pain; sleep; xyrem; must have chronic fatigue syndrome; no hypertension; no sleep apnea
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Bronchiolitis Obliterans Syndrome; Fatigue; Pain | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients were randomized and these received placebo
  Interventions: Drug: Placebo
- Sodium Oxybate (Active Comparator): Patients were randomized and these received the active drug
  Interventions: Drug: Sodium Oxybate

INTERVENTIONS:
Drug: Placebo — Subjects will be randomly assigned to either placebo or drug. The medication and the placebo come as a liquid and patients will start taking an initial dose about 30 min before they expect to sleep. If subjects awaken after less than 5 hrs of sleep, they will take a second dose. If they sleep more than 5 hrs, they will skip the second dose. We will call patients weekly to see how they are doing . If they have tolerable side effects or report significant improvement, we will maintain the dose. But if patients report no effect, the dosage will be incremented by 1 ml per week until good sleep is achieved or a predetermined maximum is reached.
  Arms: Placebo
Drug: Sodium Oxybate — Subjects will be randomly assigned to either placebo or drug. The medication and the placebo come as a liquid and patients will start taking an initial dose about 30 min before they expect to sleep. If subjects awaken after less than 5 hrs of sleep, they will take a second dose. If they sleep more than 5 hrs, they will skip the second dose. We will call patients weekly to see how they are doing . If they have tolerable side effects or report significant improvement, we will maintain the dose. But if patients report no effect, the dosage will be incremented by 1 ml per week until good sleep is achieved or a predetermined maximum is reached.
  Other Names: Xyrem
  Arms: Sodium Oxybate

SUMMARY:
Chronic fatigue syndrome is a disabling illness for which there is no specific treatment. As a group, CFS patients have disturbed sleep with frequent arousals and the sense of not having slept upon awakening. Xyrem (Sodium oxybate) is known to improve deep sleep and so may reduce the sleep disturbances of CFS leading to better sleep with less fatigue. Its ability to produce the rapid onset of deep sleep is a reason it became a street drug, but its availability is currently limited via distribution through a single centralized pharmacy. Xyrem has been successfully used based on results from a study on patients with fibromyalgia (FM), an ailment closely resembling CFS. However, in that study, the researchers provided no information as to whether patients had FM alone or FM plus CFS. Thus, it is not clear from this study just which patient may be helped. I have prescribed Xyrem for patients who have both FM and CFS with good results. In this study, funded by the company that makes Xyrem, I propose testing the drug's efficacy on patients with CFS alone - that is, they do not have fibromyalgia.

Volunteers for this study will complete paper and pencil questionnaires about their symptoms as well as a computerized test to assess their degree of brain fog. They will then be randomly assigned to one of two groups, placebo or drug. Volunteers will not know what group they are in until the end of the study. Only the drug group will receive the medication. The placebo group will receive a substance that looks identical to the real medicine but with no active ingredients. The medication comes as a liquid and patients will start taking an initial dose about 30 min before they expect to sleep. If subjects awaken after less than 5 hrs of sleep, they will take a second dose. If they sleep more than 5 hrs, they will be told to skip taking the second dose. We will call patients weekly to see how they are doing on the "drug." If they have tolerable side effects or report significant improvement, we will maintain the dose. But if patients report no effect of treatment, the dosage will be incremented by 1 ml per week until good sleep is achieved or a predetermined maximum is reached.

DETAILED DESCRIPTION:
Medically unexplained fatigue occurs in about 5% of the population with 10% of that number fulfilling formal case definitions for chronic fatigue syndrome1. Medically unexplained fatigue is a major problem for both patient and practitioner - for both because there is no effective FDA-approved treatment for the symptom. One major problem for these patients is unrefreshing sleep. Formal sleep studies show reduced total sleep time and reduced sleep efficiency compared to controls.2;3 We are currently in the early stages of an NIH-funded grant designed to study cytokines during sleep. Preliminary results support awake time for patients relative to controls, producing a decreased sleep efficiency. These data lead to our working hypothesis that the problem of severe daytime fatigue is due to a previously unappreciated form of sleep pathology related to sleep fragmentation.

Patients with medically unexplained pain also complain of disturbed sleep. Sodium oxybate has been tested on patients with this complaint who fulfill a formal case definition for fibromyalgia and has found to reduce symptoms and improve sleep quality.4 Specifically, six of 7 pain/fatigue scores (overall pain, pain at rest, pain during movement, end of day fatigue, overall fatigue, and morning fatigue) were relieved by 29% to 33% with sodium oxybate, compared with 6% to 10% relief with placebo (p < 0.005). Alpha intrusion indicative of disturbed sleep, sleep latency, and rapid-eye-movement sleep were significantly decreased, while slow-wave (stage 3/4) sleep was significantly increased, compared with placebo (p < 0.005). Two of the 5 subjective sleep related variables were significantly different from placebo: morning alertness (improved by 18% with sodium oxybate, compared with 2% for placebo; p = 0.0033) and quality of sleep (improved by 33% and 10%, respectively; p = 0.0003).

Importantly, approximately 40% of patients in my study group fulfill case definitions simultaneously for CFS and FM. Since we do not know if patients in either sodium oxybate treatment trial had CFS, we cannot be sure whether efficacy was specific for FM or instead may have occurred due to the fact that a large representation of CFS had occurred.

An unpublished Phase II randomized double-blind placebo controlled trial in FM, done by Jon Russell and colleagues in Dallas and presented at the 2005 meeting of the American College of Rheumatology, reported substantial symptom improvement with statistically significant benefits in self reported pain scales and patient global impression of improvement at both doses of sodium oxybate tested compared with placebo [4.5g [9ml] total dose per night; p=0.005 and 6g [12 ml], p=0.048]. Improvement in outcome variables was 34.5% at the 4.5g and 27.3% at the 6g compared to 12.5% in the placebo group.

I have prescribed sodium oxybate in my own practice for patients who have both CFS and FM with good results. Anecdotally, patients reporting less pain also reported better quality sleep and less fatigue upon awakening. This has led me to hypothesize that sodium oxybate will reduce fatigue in patients with CFS alone (i.e., without also having FM).

To test this hypothesis, I propose doing a double blind, placebo controlled trial of sodium oxybate in 30 patients who fulfill a formal case definition for chronic fatigue syndrome and who do not also have FM.

ELIGIBILITY:
Inclusion Criteria:

• I have CFS

Exclusion Criteria:

* I do not meet the above criteria
* I have a lifelong history of fatigue
* I have Fibromyalgia
* I have hypertension
* I am pregnant or breastfeeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Natelson, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ - Pain & Fatigue Study Center, ADMC 1618, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Xyrem: Volunteers will complete questionnaires about their symptoms. They will be randomly assigned to one of two groups, placebo or drug. Volunteers will know what group they are in at end of the study. Only the drug group will receive the medication. The placebo group will receive a substance that looks like the real medicine but with no active ingredients. The medication comes as a liquid and patients will start taking an initial dose about 30 min before they expect to sleep. If subjects awaken after less than 5 hrs of sleep, they will take a second dose. If they sleep more than 5 hrs, they will skip the second dose. We will call patients weekly to see how they are doing . If they have tolerable side effects or report significant improvement, we will maintain the dose. But if patients report no effect, the dosage will be incremented by 1 ml per week until good sleep is achieved or a predeterm
- Xyrem: Xyrem: Same as for Placebo
Period: Overall Study
Arm/Group | Placebo | Xyrem
Started | 7 | 10
Completed | 6 | 5
Not Completed | 1 | 5
Not completed — Adverse Event | 1 | 5

BASELINE CHARACTERISTICS:
Population: No info available
Groups:
- Placebo: Xyrem: Volunteers will complete questionnaires about their symptoms and a computerized test to assess their degree of brain fog. They will be randomly assigned to one of two groups, placebo or drug. Volunteers will know what group they are in at end of the study. Only the drug group will receive the medication. The placebo group will receive a substance that looks like the real medicine but with no active ingredients. The medication comes as a liquid and patients will start taking an initial dose about 30 min before they expect to sleep. If subjects awaken after less than 5 hrs of sleep, they will take a second dose. If they sleep more than 5 hrs, they will skip the second dose. We will call patients weekly to see how they are doing . If they have tolerable side effects or report significant improvement, we will maintain the dose. But if patients report no effect, the dosage will be incremented by 1 ml per week until good sleep is achieved or a predeterm
- Total: Total of all reporting groups
Arm/Group | Placebo | Xyrem | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17
Initial illness severity rating [Number; unit: participants] | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Global Assessment of Change
Description: A count was made of subject responses on a Patient Assessment of Change questionnaire where scores went from +2 [much better] thru 0 [no change] to -2 [much worse]
Time Frame: 6 weeks
Population: Had we completed the study, the analysis would have been a comparison of counts of those reporting being very much improved across the two treatment conditions
Measure: Number; unit: participants
Groups:
- Placebo; Drug Treated: Xyrem: Volunteers will complete questionnaires. They will be randomly assigned to one of two groups, placebo or drug. Volunteers will know what group they are in at end of the study. Only the drug group will receive the medication. The placebo group will receive a substance that looks like the real medicine but with no active ingredients. The medication comes as a liquid and patients will start taking an initial dose about 30 min before they expect to sleep. If subjects awaken after less than 5 hrs of sleep, they will take a second dose. If they sleep more than 5 hrs, they will skip the second dose. We will call patients weekly to see how they are doing . If they have tolerable side effects or report significant improvement, we will maintain the dose. But if patients report no effect, the dosage will be incremented by 1 ml per week until good sleep is achieved.
Arm/Group | Placebo | Drug Treated
Number analyzed (Participants) | 6 | 5
participants | 6 | 5
Statistical Analysis 1: Comparison: Placebo vs Drug Treated; Null Hypothesis = drug-treated would have a higher global impression of change than placebo treated; Test type: Superiority or Other; p < 0.04, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Self Reported Assessment of Sleep
Description: Subjects were asked to provide their input as to the quality of their sleep over the past week
Time Frame: Assessed at week 6
Population: While data were collected, these data were never analyzed because the study was terminated prematurely by the sponsor and were lost when PI moved from UMDNJ to Beth Israel in NYC in 2008.
Arm/Group | Placebo | Xyrem
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Xyrem
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 1/7 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | Xyrem (N=10)
Gastric upset (Gastrointestinal disorders) | 1 | 5

LIMITATIONS AND CAVEATS:
Too few subjects to get any definitive data. Based on the preliminary data analysis done with available subjects, we infer that had we completed the study, we might have found a significant effect for drug treated over placebo treated subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No